CLINICAL TRIAL: NCT05339100
Title: A Multicenter, Randomized, Open-label, Parallel Phase 1 Comparability Study of Anifrolumab Administered Using Accessorized Pre-Filled Syringe (APFS) or Autoinjector (AI) in Healthy Volunteers
Brief Title: Accessorized Pre-Filled Syringe to Autoinjector Pharmacokinetic Bridging Study in Anifrolumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D3465C00002; 2021-004896-14 (EudraCT Number)
Record Dates: First submitted 2022-03-07; First posted 2022-04-21 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Healthy Participants Study
Keywords: Monoclonal Antibody; Anifrolumab; Anifrolumab administered using autoinjector; Anifrolumab administered using accessorized pre-filled syringe
MeSH Terms: interventions — anifrolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anifrolumab administered using AI (Experimental): Randomized participants will receive a single SC dose of anifrolumab via AI.
  Interventions: Drug: Anifrolumab; Device: Autoinjector
- Anifrolumab administered using APFS (Active Comparator): Randomized participants will receive a single SC dose of anifrolumab via APFS.
  Interventions: Drug: Anifrolumab; Device: Accessorized Pre-Filled Syringe

INTERVENTIONS:
Drug: Anifrolumab — Participants will receive SC doses anifrolumab via AI or APFS.
Device: Autoinjector — Autoinjector will be use to administer single SC dose of anifrolumab.
  Arms: Anifrolumab administered using AI
Device: Accessorized Pre-Filled Syringe — Accessorized Pre-filled syringe will be use to administer single SC dose of anifrolumab.
  Arms: Anifrolumab administered using APFS

SUMMARY:
This study will be conducted to compare the pharmacokinetic (PK) exposure after a single SC dose of anifrolumab administered using an AI with the PK exposure after a single subcutaneous (SC) dose of anifrolumab administered using APFS in healthy male and female volunteers.

DETAILED DESCRIPTION:
This will be a multicenter, randomized, open-label, parallel group Phase 1 study.

After meeting the eligibility criteria, all eligible participants will be randomized 1:1:1:1:1:1 to a device group (APFS or AI) for an anatomical injection site as defined in the protocol. Randomization will be stratified by protocol defined body weight categories and clinical unit.

The study will comprise:

* A Screening Period up to 28 days.
* One treatment period during which eligible participants will be admitted to the Clinical Unit on Day -1 to reassess their eligibility. Participants who meet eligibility criteria will be randomized to receive a single subcutaneous (SC) dose of anifrolumab by either APFS or AI device on Day 1. Participants will be discharged on Day 3.
* The participants will return to the center for Follow-up Visits on Days 6, 8, 12, 15, 22, 29, and 43.
* A final Follow-up Visit on Day 57.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants (childbearing and non-childbearing potential) aged 18 - 55 years (inclusive) at Screening with suitable veins for cannulation or repeated venipuncture at screening.
* Female participants of childbearing potential must have a negative pregnancy test at Screening.
* Female participants of childbearing and non-childbearing potential and male participants must adhere to the contraception methods.
* Have a body mass index between 18.5 and 30 kg/m^2 inclusive and weigh at least 50 kg and no more than 110 kg inclusive at Screening.
* Participants must have immunity against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), either by having recovered from a SARS-CoV-2 infection (should have recovered from infection at least 6 weeks before Screening Visit as confirmed by a COVID-19 test) or fully vaccinated against SARS CoV-2 with vaccines approved in the local region (should have received the final vaccine dose at least 2 weeks before Screening Visit).
* Participant should meet all of following tuberculosis (TB) criteria:

  1. No signs or symptoms of active TB prior to or during any Screening Visit.
  2. No medical history or past physical examinations suggestive of active TB.
  3. No recent contact with a person with active TB OR if there has been such contact, referral to a physician specializing in TB to undergo additional evaluation prior to randomization (documented comprehensively in source), and, if warranted, receipt of appropriate treatment for latent TB at or before the first administration of investigational product.
  4. No history of latent TB prior to initial Screening visit, with the exception of latent TB with documented completion of appropriate treatment.
* Negative result for an Interferon-gamma (IFN-γ) release assay (IGRA) (eg QuantiFERON-TB Gold [QFT-G] test) test for TB at screening.

Exclusion Criteria:

* Lactating or pregnant females or females who intend to become pregnant or begin breastfeeding anytime from initiation of Screening until 1 month after the final Follow-up Visit.
* History or presence of hepatic or renal diseases known to interfere with the PK of anifrolumab.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the administration of study intervention, as judged by the Investigator.
* Any clinically significant abnormalities in in clinical chemistry, hematology, or urinalysis results, at Screening and/or admission to the Clinical Unit.
* Any clinically significant abnormal findings in vital signs at Screening and/or admission to the Clinical Unit.
* Any clinically significant abnormalities on 12-lead electrocardiogram at Screening, as judged by the Investigator.
* Any positive result on Screening for serum hepatitis B surface antigen OR anti-HBc antibody, hepatitis C antibody, and Human immunodeficiency virus antibody.
* Opportunistic infection requiring hospitalization or IV antimicrobial treatment within 3 years of randomization.
* Clinically significant chronic infection (eg, osteomyelitis, bronchiectasis, etc.) within 8 weeks prior to signing the informed consent form (ICF).
* Any infection requiring hospitalization or treatment with IV anti-infective medications not completed at least 4 weeks prior to signing the ICF.
* Any infection requiring oral anti-infective medications (including antivirals) within 2 weeks prior to Day 1.
* History of severe Coronavirus Disease 2019 (COVID-19) infection requiring hospitalization within the last 12 months prior to Screening, or clinical history compatible with Long COVID 19 (symptoms beyond 12 weeks of acute infection), as judged by the Investigator.
* COVID-19 infection before or during Screening and/or admission confirmed by a COVID 19 test (at the London Clinical Unit, participants will have a PCR test on Day -2 only. Additional testing may be performed as required at the discretion of the investigator.
* Known or suspected history of drug abuse, as judged by the Investigator.
* Positive screen for drugs of abuse or cotinine at Screening or on admission to the Clinical Unit or positive screen for alcohol at Screening or on admission to the Clinical Unit.
* Participation in another clinical trial, or has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the administration of SI in this study. The period of exclusion begins 3 months after the final dose or 5 half-lives, whichever is the longest.
* Plasma donation within 1 month of Screening or any blood donation/loss more than 500 mL during the 3 months prior to Screening.
* A known history of allergy or reaction to any component of the IP formulation or history of anaphylaxis to any human gamma globulin therapy.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to Screening.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the administration of SI.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the Investigator. Excessive intake of alcohol defined as the regular consumption of more than 24 g of alcohol per day for men or 12 g of alcohol per day for women (for the London unit: regularly consuming >21 units of alcohol per week for males or >14 units of alcohol per week for females).
* Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate) as judged by the Investigator. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day (eg, >5 cups of coffee) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the investigational site.
* Participants who have previously received anifrolumab.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Area under serum concentration-time curve from time zero extrapolated to infinity (AUCinf) | Up to Day 57
  Evaluation of AUCinf following single SC administration of anifrolumab by AI is comparable to the AUCinf following single SC administration of anifrolumab using APFS will be done.
Area under serum concentration-time curve from time zero to last quantifiable concentration (AUClast) | Up to Day 57
  Evaluation of AUClast following single SC administration of anifrolumab by AI is comparable to the AUClast following single SC administration of anifrolumab using APFS will be done.
Maximum observed serum (peak) drug concentration (Cmax) | Up to Day 57
  Evaluation of Cmax following single SC administration of anifrolumab by AI is comparable to the Cmax following single SC administration of anifrolumab using APFS will be done.

SECONDARY OUTCOMES:
Time to reach peak or maximum observed concentration (tmax) | Day 1 to Day 57
  Evaluation of the tmax of anifrolumab administered to various anatomical injection sites and in healthy participants within different body weight ranges.
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t1/2λz) | Day 1 to Day 57
  Evaluation of the t1/2λz of anifrolumab administered to various anatomical injection sites and in healthy participants within different body weight ranges will be done.
Mean residence time of the unchanged drug in the systemic circulation from zero to infinity (MRT) | Day 1 to Day 57
  Evaluation of the MRT of anifrolumab administered to various anatomical injection sites and in healthy participants within different body weight ranges will be done.
Apparent total body clearance of drug after extravascular administration (CL/F) | Day 1 to Day 57
  Evaluation of the CL/F of anifrolumab administered to various anatomical injection sites and in healthy participants within different body weight ranges will be done.
Apparent volume of distribution following extravascular administration (based on terminal phase) (Vz/F) | Day 1 to Day 57
  Evaluation of the Vz/F of anifrolumab administered to various anatomical injection sites and in healthy participants within different body weight ranges will be done.
Time of last quantifiable concentration (tlast) | Day 1 to Day 57
  Evaluation of the tlast of anifrolumab administered to various anatomical injection sites and in healthy participants within different body weight ranges will be done.
Number of participants with positive Anti-drug antibodies (ADA) | Day 1, 29 and 57
  Evaluation of the immunogenicity of anifrolumab delivered by AI or APFS will be done.
Number of participants with adverse events and serious adverse events | Screening period (Day -28 to Day-2) through follow-up visit (Day 57) and evaluation of injection site reaction (Days 1 to 3)
  Evaluation of safety and tolerability of AI- vs APFS-administered anifrolumab will be done.

CONTACTS AND LOCATIONS:
Locations (3):
- Research Site, Brooklyn, Maryland, United States
- Research Site, Berlin, Germany
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patientlevel data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home